CLINICAL TRIAL: NCT01929889
Title: An Exploratory Study to Assess the Effects of Fanapt® on Social Cognitive Performance
Brief Title: Assessing the Effects of Fanapt® on Social Cognition in Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Northwestern University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, John Csernansky, Lizzie Gilman Professor and Chairman, Department of Psychiatry and Behavioral Sciences, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIL0522DUS03T
Record Dates: First submitted 2013-08-19; First posted 2013-08-28 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; iloperidone; Fanapt; social cognition; cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — iloperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iloperidone (Experimental): Patients currently taking an antipsychotic medication other than Fanapt® will switch from their current medicine to Fanapt® in a cross-titration at a rate that is determined by the study physician. Treatment with iloperidone will be initiated and dosage will increase until the subject has achieved clinical stability, or has achieved the maximum dose, or 8 weeks have elapsed. Subjects who do not achieve clinical stability (as defined in the inclusion criteria) for the final 2 weeks in this 8-week period at the maximum dose of iloperidone will be discontinued from the study. If patients achieve stabilization, the lowest effective dose will be maintained. Subjects who have achieved clinical stability will then enter the 12-week treatment phase of the study.
  Interventions: Drug: Iloperidone

INTERVENTIONS:
Drug: Iloperidone — Patients in this study will be treated with Fanapt® (iloperidone). They will begin a standardized up-titration starting with a dose of 2 mg daily. Dose increases will continue until the subject has achieved clinical stability, has achieved the maximum dose of 24 mg/day, or until 8 weeks have elapsed. Once clinical stability has been achieved, the patient will continue into the treatment phase. If clinical stability is not achieved after 8 weeks, the patient will be excluded from the study.
  Other Names: Fanapt

SUMMARY:
The study looks at whether treatment with iloperidone (Fanapt) is associated with improvements in social cognition in individuals who have been recently diagnosed with schizophrenia or schizoaffective disorder. Social cognition (the ability to understand your feelings and the feelings of others) is closely related to functional outcomes, including communication, empathy, and emotional recognition.

DETAILED DESCRIPTION:
Schizophrenia is a disabling disease that affects about 1% of the population and is one of the leading causes of psychiatric disability. Striking early in life, schizophrenia interferes with work, relationships, and independence. Despite the billions of dollars spent annually in the direct and indirect costs of this disease, there are few treatment options that restore functionality. Lately, cognition has emerged as a target for interventions, since a patient's cognitive status is one of the most reliable predictors of functional outcome, and yet treatments for improving cognition have delivered only modest results. This study will attempt to evaluate the efficacy of Fanapt® (iloperidone) on social cognition, which consists of factors such as empathy, social perception, and emotional recognition, and may be more meaningfully tied to functional outcome than cognition in general.

This study will assess social cognition in people with schizophrenia or schizoaffective disorder who have newly begun taking Fanapt® (iloperidone), a new antipsychotic with mixed dopamine and serotonin antagonism. Standard measures of psychopathology and social cognition will be collected at baseline and then again at 12 weeks after becoming stable on the medication, by raters who are blind to the length of a subject's participation in the study. We predict that social cognition will improve with treatment with Fanapt®. This study has relatively few risks, including no risks beyond exposure to the study medication and the collection of safety data and psychometric data. The potential benefits outweigh the risks, with the main benefit being an ability to describe an improvement in cognitive performance that is believed to relate directly to real-world functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent
* Male and female patients 18-55 years old
* DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder.
* Less than 5-year treatment history for schizophrenia or schizoaffective disorder.
* Clinically stable for the last 2 weeks of the Fanapt® screening and stabilization phases.
* Sufficiently stable overall health.
* Women who can become pregnant must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study

Exclusion Criteria:

* People unable to give informed consent
* Baseline performance of 95% or higher on the cognitive empathy assessment
* Pregnant and lactating women
* A positive test for Hepatitis C antibody with concurrent evidence of impaired hepatic function
* Subjects with a history of medical conditions which would pose a risk to the patient if they were to participate in the study or that might confound the results of the study
* Known hypersensitivity to Fanapt® or any components in its formulation
* History of organic brain disorder
* History of autism, pervasive developmental disability, mental retardation, or other cognitive disorder that could potentially confound cognitive testing
* History of any medical condition that would confound the presentation or treatment of schizophrenia or schizoaffective disorder, or significantly increase the risk associated with the proposed treatment protocol
* History of QTc prolongation, cardiac arrhythmias, or family history of sudden cardiac death
* Patients taking strong inhibitors of CYP2D6 (fluoxetine, paroxetine, etc.) or CYP3A4 (ketoconazole, itraconazole, cimetidine, cyclosporine, etc.) or other medications that interact significantly with iloperidone
* Patients who have met DSM-IV-TR criteria for current alcohol or substance dependence within the last six months or DSM-IV-TR criteria for alcohol or substance abuse within the last month
* Patients regularly taking any medication that is known to interfere with performance on cognitive and social cognitive tasks, such as anticholinergics and benzodiazepines. Occasional benzodiazepine use may be permitted if subject can safely refrain from use for at least 24 hours prior to study visits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Csernansky, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Barch DM, Smith E. The cognitive neuroscience of working memory: relevance to CNTRICS and schizophrenia. Biol Psychiatry. 2008 Jul 1;64(1):11-7. doi: 10.1016/j.biopsych.2008.03.003. Epub 2008 Apr 8. PMID 18400207
- [Background] Bell M, Tsang HW, Greig TC, Bryson GJ. Neurocognition, social cognition, perceived social discomfort, and vocational outcomes in schizophrenia. Schizophr Bull. 2009 Jul;35(4):738-47. doi: 10.1093/schbul/sbm169. Epub 2008 Jan 31. PMID 18245058
- [Background] Bell MD, Zito W, Greig T, Wexler BE. Neurocognitive enhancement therapy with vocational services: work outcomes at two-year follow-up. Schizophr Res. 2008 Oct;105(1-3):18-29. doi: 10.1016/j.schres.2008.06.026. Epub 2008 Aug 19. PMID 18715755
- [Background] Bellack AS, Schooler NR, Marder SR, Kane JM, Brown CH, Yang Y. Do clozapine and risperidone affect social competence and problem solving? Am J Psychiatry. 2004 Feb;161(2):364-7. doi: 10.1176/appi.ajp.161.2.364. PMID 14754789
- [Background] Brekke J, Kay DD, Lee KS, Green MF. Biosocial pathways to functional outcome in schizophrenia. Schizophr Res. 2005 Dec 15;80(2-3):213-25. doi: 10.1016/j.schres.2005.07.008. Epub 2005 Aug 30. PMID 16137859
- [Background] Brune M. Emotion recognition, 'theory of mind,' and social behavior in schizophrenia. Psychiatry Res. 2005 Feb 28;133(2-3):135-47. doi: 10.1016/j.psychres.2004.10.007. PMID 15740990
- [Background] Combs DR, Adams SD, Penn DL, Roberts D, Tiegreen J, Stem P. Social Cognition and Interaction Training (SCIT) for inpatients with schizophrenia spectrum disorders: preliminary findings. Schizophr Res. 2007 Mar;91(1-3):112-6. doi: 10.1016/j.schres.2006.12.010. Epub 2007 Feb 12. PMID 17293083
- [Background] Derntl B, Finkelmeyer A, Toygar TK, Hulsmann A, Schneider F, Falkenberg DI, Habel U. Generalized deficit in all core components of empathy in schizophrenia. Schizophr Res. 2009 Mar;108(1-3):197-206. doi: 10.1016/j.schres.2008.11.009. Epub 2008 Dec 16. PMID 19087898
- [Background] Glynn SM, Cohen AN, Dixon LB, Niv N. The potential impact of the recovery movement on family interventions for schizophrenia: opportunities and obstacles. Schizophr Bull. 2006 Jul;32(3):451-63. doi: 10.1093/schbul/sbj066. Epub 2006 Mar 8. PMID 16525087
- [Background] Harvey PD, Penn D. Social cognition: the key factor predicting social outcome in people with schizophrenia? Psychiatry (Edgmont). 2010 Feb;7(2):41-4. PMID 20376275
- [Background] Kane JM, Lauriello J, Laska E, Di Marino M, Wolfgang CD. Long-term efficacy and safety of iloperidone: results from 3 clinical trials for the treatment of schizophrenia. J Clin Psychopharmacol. 2008 Apr;28(2 Suppl 1):S29-35. doi: 10.1097/JCP.0b013e318169cca7. PMID 18334910
- [Background] Penn DL, Roberts DL, Combs D, Sterne A. Best practices: The development of the Social Cognition and Interaction Training program for schizophrenia spectrum disorders. Psychiatr Serv. 2007 Apr;58(4):449-51. doi: 10.1176/ps.2007.58.4.449. PMID 17412842
- [Background] Roberts DL, Penn DL, Labate D, Margolis SA, Sterne A. Transportability and feasibility of Social Cognition And Interaction Training (SCIT) in community settings. Behav Cogn Psychother. 2010 Jan;38(1):35-47. doi: 10.1017/S1352465809990464. Epub 2009 Oct 27. PMID 19857363
- [Background] Wolwer W, Frommann N, Halfmann S, Piaszek A, Streit M, Gaebel W. Remediation of impairments in facial affect recognition in schizophrenia: efficacy and specificity of a new training program. Schizophr Res. 2005 Dec 15;80(2-3):295-303. doi: 10.1016/j.schres.2005.07.018. Epub 2005 Aug 24. PMID 16125367
- [Result] Andreasen NC, Arndt S, Alliger R, Miller D, Flaum M. Symptoms of schizophrenia. Methods, meanings, and mechanisms. Arch Gen Psychiatry. 1995 May;52(5):341-51. doi: 10.1001/archpsyc.1995.03950170015003. PMID 7726714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study target enrollment goal was 20 completed subjects.
Pre-assignment Details: 19 subjects were consented and completed the study screening visit.11 subjects did not start on the treatment after signing the consent form. The most common reason for early termination was disagreement between the subjects' self-reported diagnosis and the diagnosis obtained by the research psychiatrist.
Groups:
- A Single Arm, Open Label, Exploratory Study: This is a single arm, open label, exploratory study to examine effects of Fanapt (iloperadone) on social cognition. Patients currently taking an antipsychotic medication other than Fanapt® will switch from their current medicine to Fanapt® in a cross-titration at a rate that is determined by the study physician. Treatment with iloperidone will be initiated and dosage will increase until the subject has achieved clinical stability, or has achieved the maximum dose, or 8 weeks have elapsed. Subjects who do not achieve clinical stability (as defined in the inclusion criteria) for the final 2 weeks in this 8-week period at the maximum dose of iloperidone will be discontinued from the study. If patients achieve stabilization, the lowest effective dose will be maintained. Subjects who have achieved clinical stability will then enter the 12-week treatment phase of the study.
Period: Overall Study
Arm/Group | A Single Arm, Open Label, Exploratory Study
Started | 8 (Target enrollment goal was 20 completed subjects.)
Completed | 3 (3 subjects completed the study.)
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Iloperidone
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Social Cognition at 12 Weeks
Description: Facial Affect Perception Test that assesses the ability to accurately recognize facially expressed emotions as published by Smith et al 2014; Derntl et al., 2009. This scale ranges from 0-100 percent with a total of 30 trials. We examined the percent correct as the total number of correct responses divided by the total number of completed trials. There were no subscales. 100% accurate is the best outcome and 0% accurate is the worst outcome.
  Cognitive Empathy Test that assesses the ability to accurately determine the emotional expression of another person as depicted in a static image of a social interaction as published by Smith et al 2014; Derntl et al., 2009. This scale ranges from 0-100 percent with a total of 60 trials. We examined the percent correct as the total number of correct responses divided by the total number of completed trials. There were no subscales. 100% accurate is the best outcome and 0% accurate is the worst outcome.
Time Frame: baseline and twelve weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iloperidone
Number analyzed (Participants) | 3
units on a scale
  Facial Affect Perception Test | 0 (3.742)
  Cognitive Empathy Test | -3.333 (6.807)

ADVERSE EVENTS:
Time Frame: Adverse events were systematically collected throughout the study.
Arm/Group | Iloperidone
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iloperidone (N=8)
Hospitalization (Psychiatric disorders) | 3 (3) — Emergent suicidal ideation (n.b., no suicide attempt was made). The subject was admitted to hospital.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iloperidone (N=8)
Abdominal pain (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The most common reason for early termination was disagreement between the subjects' self-reported diagnosis and the diagnosis obtained by the research psychiatrist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes